CLINICAL TRIAL: NCT00610948
Title: A Sequential Phase I Study Of The Combination Of Everolimus (Rad001) With 5-Fu/Lv (De Gramont), Folfox6, And Folfox6/Panitumumab In Patients With Refractory Solid Malignancies
Brief Title: Everolimus, Fluorouracil, Leucovorin, Panitumumab, and Oxaliplatin in Treating Patients With Tumors That Did Not Respond to Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0621; P30CA016086 (NIH); CDR0000584276 (Other: PDQ number)
Record Dates: First submitted 2008-02-07; First posted 2008-02-08 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Panitumumab; Everolimus; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Patients receive oral everolimus once daily on days 1-28. Patients also receive leucovorin calcium IV followed by fluorouracil IV continuously over 46 hours beginning on day 1. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: everolimus; Drug: fluorouracil; Drug: leucovorin calcium
- Group 2 (Experimental): Patients receive oral everolimus once daily on days 1-28 and panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: panitumumab; Drug: everolimus
- Group 3 (Experimental): Patients receive oral everolimus once daily on days 1-28, leucovorin calcium IV followed by fluorouracil IV continuously over 46 hours beginning on day 1, and oxaliplatin IV over 2-4 hours on day 1. Some patients may also receive panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: panitumumab; Drug: everolimus; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Biological: panitumumab — Given IV
  Other Names: Vectibix
  Arms: Group 2; Group 3
Drug: everolimus — Given orally
  Other Names: Afinitor
Drug: fluorouracil — Given IV
  Other Names: 5FU
  Arms: Group 1; Group 3
Drug: leucovorin calcium — Given IV
  Arms: Group 1; Group 3
Drug: oxaliplatin — Given IV
  Other Names: Eloxatin
  Arms: Group 3

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as fluorouracil, leucovorin, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving everolimus together with combination chemotherapy and/or panitumumab may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of everolimus when given together with fluorouracil, leucovorin, panitumumab, and oxaliplatin in treating patients with solid tumors that did not respond to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of everolimus in combination with sequential fluorouracil (5-FU) and leucovorin calcium, panitumumab, modified 5-FU, leucovorin calcium, and oxaliplatin (mFOLFOX6), and mFOLFOX6 with panitumumab in patients with refractory solid tumors.

Secondary

* To determine the adverse event profile of these regimens.
* To correlate response with S6-phosphorylation and AKT-phosphorylation in available archived tumor samples.
* To evaluate preliminary evidence of antitumor activity of these regimens using RECIST criteria for a subset of patients with measurable disease.

OUTLINE: This is a dose-escalation study. Cohorts of patients are enrolled into treatment groups 1 or 2. If a final cohort of patients is reached in groups 1 and/or 2, additional cohorts of patients are enrolled into treatment group 3.

* Group 1: Patients receive oral everolimus once daily on days 1-28. Patients also receive leucovorin calcium IV followed by fluorouracil IV continuously over 46 hours beginning on day 1. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
* Group 2: Patients receive oral everolimus once daily on days 1-28 and panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
* Group 3: Patients receive oral everolimus once daily on days 1-28, leucovorin calcium IV followed by fluorouracil IV continuously over 46 hours beginning on day 1, and oxaliplatin IV over 2-4 hours on day 1. Some patients may also receive panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Archived tumor samples are assessed for phospho-AKT, phospho-S6K, and phospho-S6 by immunohistochemistry.

After completion of study treatment, patients are followed every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumor

  * Advanced or unresectable disease
* No standard therapeutic option available
* Evaluable disease (according to RECIST criteria) that has not been previously irradiated

  * Prior radiotherapy to the marker lesion(s) allowed provided there is evidence of progression since radiotherapy
* Brain metastases allowed provided the following criteria are met:

  * CNS-directed treatment was given and was completed > 3 months ago
  * CNS disease has been clinically and radiographically stable for ≥ 8 weeks

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/µL
* Platelet count ≥ 100,000/µL
* Creatinine clearance ≥ 60 mL/min
* Total bilirubin ≤ 1.2 mg/dL
* Transaminases ≤ 5 times upper limit of normal (ULN)
* Magnesium ≥ lower limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 24 weeks (females) or for 4 weeks (males) after completion of study therapy
* Willing to avoid pregnancy for 3 months after completion of study therapy
* No neuropathy ≥ grade 2
* No concurrent life-threatening acute medical illness
* No impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* No active bleeding diathesis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior major surgery, radiotherapy (including radiotherapy involving the abdomen or spine), chemotherapy, or other systemic anticancer therapy and recovered
* At least 4 weeks since prior investigational drugs
* No concurrent CYP3A4 inducers or inhibitors that cannot be substituted by a different agent
* No concurrent oral anti-vitamin K medication (except for low-dose warfarin)
* No concurrent colony stimulating factors during the first course of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-03; Primary Completion 2013-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of everolimus in combination with sequential fluorouracil (5-FU) and leucovorin calcium, panitumumab, modified 5-FU, leucovorin calcium, and oxaliplatin (mFOLFOX6), and mFOLFOX6 with panitumumab | after the first 28 day cycle
  Patients will be assessed for toxicity at the commencement of each cycle
Toxicity as assessed by CTC version 3.0 at the beginning of each treatment course | first 28 day cycle
  Dose Limiting Toxicities (DLT) are defined during the first cycle (28 days).
Tumor response | Every 8 weeks during treatment
  Tumor response will be assessed by RECIST criteria
Correlation of response with S6-phosphorylation and AKT-phosphorylation in archived tumor samples | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Autumn McRee, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] McRee AJ, Davies JM, Sanoff HG, Goldberg RM, Bernard S, Dees EC, Keller K, Ivanova A, O'Neil BH. A phase I trial of everolimus in combination with 5-FU/LV, mFOLFOX6 and mFOLFOX6 plus panitumumab in patients with refractory solid tumors. Cancer Chemother Pharmacol. 2014 Jul;74(1):117-23. doi: 10.1007/s00280-014-2474-0. Epub 2014 May 13. PMID 24819684
- See also: web address for the National Cancer Institute (NCI) — http://www.cancer.gov
- See also: web address for the Lineberger Comprehensive Cancer Center, UNC — http://www.unclineberger.org